CLINICAL TRIAL: NCT07108920
Title: Analysis of Balance Disorders After Botulinum Toxin Treatment in the Rectus Femoris in Patients With a Stiff Knee Gait: What About the Risk of Falls?
Brief Title: Analysis of Balance Disorders After Botulinum Toxin Treatment in the Rectus Femoris in Patients With a Stiff Knee Gait
Acronym: FEMFALLTOX
Status: Recruiting | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-07-FEMFALLTOX
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-07

CONDITIONS: Botulinum Toxin Injection; Stiff Knee Gait; Fall Risk; Rectus Femoris Muscle; Botox Injection; Spasticity With Multiple Sclerosis
Keywords: Botulinum toxin injection; Rectus femoris; Balance troubles; Fall risk analysis; Stiff knee gait patients.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with botulinum toxin injection in the rectus femoris.
  Interventions: Other: Functional clinical tests

INTERVENTIONS:
Other: Functional clinical tests — Functional clinical tests:
  * Time Up and Go test
  * Berg Balance Scale (BBS)
  * Stair climb and descent time test (SCT)
  * Number of falls via a questionnaire

SUMMARY:
Patients who suffered a stroke, cranial traumatism, medullar lesions or multiple sclerosis can present spastic muscular complications, which is particularly impairing if it concerns muscles of the leg. Muscular spastic complications of the legs can alter significantly the ability to walk because it clinically manifests itself by a stiffness of the leg, thus generating a complication called "Stif Knee Gait" (SKG). It means that the femoro-patello-tibial articulation cannot be mobilized as it should because it stays spastic instead of being mobile.

However, it remains possible to treat this kind of medical condition by using Botulinum toxin injections in the target muscle, in particular the rectus femoris (which is part of the quadriceps).

As a reminder, botulinum toxin, sold under the international common denomination "Botox®", is a neurotoxin of 150 kDa produced by the bacteria "Clostridium Botulinum" and is the most powerful natural poison known to humankind, with its DL50 between 1 and 2 nanogramms / kg in humans. This toxin works by entering the neuro-muscular synaptic junctions and by linking itself to a proteic complex called SNARE. The link between the toxin and the SNARE complex inhibits the fusion of the acetylcholinergic synaptic vesicles with the plasmic membrane of the pre-synaptic axone. The Botox® blocks the exocytosis of the acetycholin (Ach) vesicle in the inter-synaptic space at the neuro-muscular junction and blocks the nervous transmission, thus generating muscular flaccid paralysis. This kind of intoxication is caused directly by an infection by Clostridium Botulinum and is called Botulism. It manifests itself clinically by flaccid paralysis, swelling, diarrhea tiredness, respiratory failure, vomiting etc…

Despite its highly toxic properties, Botox® can be used as a therapeutic tool against number of medical conditions (strabismus, hyperhidrosis, migraines etc…) and even as a cosmetic tool (anti face-wrinkles). It can be used against spastic muscular paralysis, especially like the ones encountered in the patients of this study.

The current Standard Of Care (SOC) against SKG is to inject Botox into the rectus femoris in order to counter its spasticity. It has been shown to upgrade the walking ability of SKG patients by enhancing the leg kinetics. More precisely, it has been shown to improve the fluidity of the movement of the spastic leg in SKG patients, especially the knee flexion. However, the rectus femoris' contractility remains necessary to be able to stand up statically and to stay balanced during the walk and everyday-activity and the myorelaxant properties of Botox® may be problematic and alter the leg biomechanics despite its utility. To this day, no study has been published to compare the static and dynamic balance troubles before and after Botox injections in the rectus femoris.

The medical bibliography does not report any augmentation of the risk of fall in the case of Botox injection in the rectus femoris. However, we consider the hypothesis along which those injections can enhance the risk of fall. Therefore, we decided to conduct a monocentric, prospective observational clinical study to compare the state of the static and dynamic balance before and after Botox injections in the rectus femoris (in SKG patients) by using balance scores.

In order to complete this objective, we compared the following parameters before and after the Botox injection in SKG patients :

* Time Up and Go test(in seconds) : primary evaluation criteria
* Berg Balance Scale (BBS) : secondary evaluation criteria
* Stair climb and descent time test (SCT) : secondary evaluation criteria.
* Number of falls.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a stif knee gait (SKG) after a stroke, a post-traumatic cerebral lesion or a multiple sclerosis.
* If the patient had a stroke, it happened at least 4 month ago (before the inclusion).
* The patient has a rectus femoris spasticity ≥ 1 on the modified Ashworth Scale with the hip in extension position.
* A quadricipital muscular force ≥ 2/5 (MRC Scale)
* The patient didn't receive any botulinum toxin injection during the 3 previous months
* No modification of any anti-spastic medication during the inclusion in the actual month (Baclofène, Dantrolène).
* No neurosurgical intervention or ligamentoplasty of the quadricipital ligament during the 6 previous months.
* No recent knee traumatism with knee instability during the 6 previous weeks.

Exclusion Criteria:

* Other comorbidities invalidating the fonctionnal tests necessary for the study like : decompensated cardiac insufficiency, unstable respiratory insufficiency, coagulation troubles, neurocognitive impairments inhibiting the comprehension of isocinetical tests.
* Patient without severe phasic trouble inhibiting the patient's ability to answer the evaluation scales.
* Sensory lesions inhibiting the possibility to evaluate the walk : visual impairment, major proprioception impairment, or cerebellar ataxia.
* Severe muscular deficit : genetic myopathy, psychomotric desadaptation syndrom
* Absolute contraindication to botulinum toxin injections : urinary tract infection ; current treatment by aminoglycosidic antibiotics, severe myasthenia, urine retention in patient who can't receive a urinary catheter.
* Patient with cognitive troubles compromitting the understanding and the realization of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients consists in patients suffering from a stiff knee gait (SKG) after a stroke, a post-traumatic cerebral lesion or a multiple sclerosis, and who never underwent any neurosurgical procedure and didn't ever change their anti-spastic treatments.
  Those patients will be seen only in hospital structure (readaptation center) and never outside (liberal practice).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Time Up and Go test. | Realized only once 4 weeks after the inclusion visit.
  This examination consist in 6 steps :
  1. Sit on a chair
  2. Stand up
  3. Walk 3 meters
  4. Make a U-turn
  5. Walk back to the chair
  6. Sit back.
  The investigator mesures (with a chronometer) the time it takes for the patient to complete the test. The timer starts when the patient stands up, and stops when the patient sits back.

SECONDARY OUTCOMES:
Assessment of Berg Balance Scale test. | 4 weeks after the Botulinum toxin injection visit.
  The Berg Balance Scale tests consists in assessing the ability of the patient to perform 14 tasks :
  * 1 : to stand up of a chair without using hands
  * 2 : to stand up without support
  * 3 : To sit without support, feet on the floor

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Médecine Physique et de Réadaptation Bretegnier, Héricourt, Nord Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No